CLINICAL TRIAL: NCT04062643
Title: OBESITY ASSOCIATION WITH RECURRENT STROKE AND CARDIOVASCULAR EVENTS
Brief Title: Obesity Effect on Stroke and Cardiovascular Events
Acronym: OSR
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Emre Kumral, Ege Neurology, Ege University
Other Study IDs: 2010/101
Record Dates: First submitted 2019-08-08; First posted 2019-08-20 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Stroke, Acute
Keywords: obesity; recurrent stroke; ischemic stroke; hemorrhagic stroke; cardiovascular events; vascular death
MeSH Terms: conditions — Stroke; Obesity; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with obesity: Obesity in those with BMI ≥30 kg/m2
  Interventions: Diagnostic Test: Obesity assessment
- Patients without obesity: Normal weight was considered in the patients with BMI <30 kg/m2
  Interventions: Diagnostic Test: Obesity assessment

INTERVENTIONS:
Diagnostic Test: Obesity assessment — Body mass index (BMI (kg/m2) was calculated from measurements of weight to the nearest kg and height

SUMMARY:
The relation between obesity and stroke recurrence is still under debate. In this study it has been sought whether baseline obesity is associated with recurrent stroke and major cardiovascular events in a long-time period.

DETAILED DESCRIPTION:
Five-years follow-up data of Ege Stroke Registry for stroke recurrence and cardiovascular events regarding to obesity were analyzed. Data include age, gender, stroke severity, neuroimaging studies, cardiovascular risk factors. Within the inclusion period, all of the included patients were followed until censoring (10th of December 2011) or readmission because of recurrent stroke, cardiovascular event or death, whichever came first. The Kaplan-Meier method was used for survival analysis. Cox proportional hazard model was applied to identify predictors of recurrent vascular events.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive stroke patients.

Exclusion Criteria:

* Incomplete baseline information, other factors making them unsuitable for follow-up,undetermined stroke, subarachnoid hemorrhage.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All stroke patients enrolled in the prospective cohort registry in Egeanregion.
Sampling Method: Probability Sample
Enrollment: 9285 (Actual)
Dates: Start 2000-04 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Stroke recurrence | 5 years
  Ischemic or hemorrhagic stroke

IPD SHARING:
Plan to Share IPD: No
If the publisher will accept to share IPD, we can give permission to share IPD.